CLINICAL TRIAL: NCT01549600
Title: A Randomized, Controlled Study To Compare the Effects of 2 Types of Dietary Fiber, Psyllium and Microcrystalline Cellulose, on Glycemic Measures in Subjects With Pre-type 2 Diabetes
Brief Title: Comparison of Psyllium and Microcrystalline Cellulose on Glycemic Measures in Subjects With Impaired Fasting Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2011063
Record Dates: First submitted 2012-03-06; First posted 2012-03-09 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-04

CONDITIONS: Impaired Fasting Glucose
MeSH Terms: interventions — Psyllium; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- psyllium (Experimental): 5.1 g psyllium husk in at least 8 ounces of water
  Interventions: Dietary Supplement: psyllium
- Microcrsytalline Cellulose (Active Comparator): 1.18 g Microcrystalline Cellulose in at least 8 ounces of water, taken twice a day
  Interventions: Dietary Supplement: Microcrystalline Cellulose

INTERVENTIONS:
Dietary Supplement: psyllium — 1 level tablespoon (~ 5.1 g psyllium husk in the psyllium product) mixed with at least 8 ounces of water, taken twice daily
  Arms: psyllium
Dietary Supplement: Microcrystalline Cellulose — 1 level tablespoon (~ 1.18 g MCC in the MCC product) mixed with at least 8 ounces of water, taken twice a day
  Arms: Microcrsytalline Cellulose

SUMMARY:
The Purpose of this study is to compare the effects of 2 types of dietary fiber, psyllium and microcrystalline cellulose (MCC), on glycemic measures in subjects with impaired fasting glucose.

DETAILED DESCRIPTION:
This study will be conducted at a single study center. Approximately 40 subjects with pre-type 2 diabetes will be enrolled and randomized in this study.

This 22-week study consists of 3 periods: an 8-week treatment period (Visits 2-4), a 6-week washout period, and an 8-week treatment period (Visits 5-7).

ELIGIBILITY:
Inclusion Criteria:

* be male or female,
* at least 18 years of age
* in generally good health for the pre-type 2 diabetes population;
* if female, be postmenopausal or if of child-bearing capacity agree to use an adequate form of contraception
* have not used any psyllium containing products within the past 3 months;
* be willing to refrain from taking any psyllium containing products during the study;
* be willing to maintain a lifestyle habits for the duration of the study;
* have a fasting serum glucose of 110 - 125 mg/dL

Exclusion Criteria:

* if female, are pregnant or nursing (lactating);
* have a history of diabetes (diagnosis) or is currently taking medications for diabetes
* participated in a clinical drug study or used investigational drug during the previous 30 days;
* have symptoms and signs suggestive of significant underlying disease, or acute onset of new symptoms and signs of major organ disease, that could become unstable during the trial requiring urgent medical intervention
* have evidence of or treatment history of malignancy within the previous 5 years;
* currently alcohol dependent;
* used anti-psychotics in the previous 3 months;
* used systemic steroidal agents within the last 30 days;
* had used oral or systemic antibiotics or any over-the-counter (OTC) bactericidal medication (eg, bismuth salts) within the last 30 days;
* has been taking any medication that may affect blood glucose or GI motility (eg, calcium channel blockers, beta blockers, antimuscarinics, salicylates etc.) for less than 30 days or 5 times the half life of the drug (need to be stable on the medication);
* have evidence of immunodeficiency including subjects currently taking systemic corticosteroids or immunosuppressive drugs
* have a major psychiatric disorder, including major depression, psychoses, alcohol or substance abuse within the past 2 years;
* has a known sensitivity or allergy to any components of study products, including psyllium and aspartame (see Section 3.5.3);
* were previously screened (ie, Visit 1 procedures) for participation in this study and failed to meet entry criteria;
* have difficulty swallowing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
fasting serum glucose | 8 weeks
  mean change from baseline in fasting serum glucose at 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John McRorie, PhD, Study Director — Procter and Gamble; Mark Feinglos, MD, Principal Investigator — Duke University; Richard Surwit, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States